CLINICAL TRIAL: NCT02263313
Title: Evaluation of Endothelial ProGenitor Cell Capture Sirolimus-Eluting Stent by Optical Coherence Tomography: the COMBO Stent 36-months Clinical End-point Extension Study (EGO-COMBO Clinical End-point Extension Study Beyond 36 Months)
Brief Title: EGO-COMBO Clinical End-point Extension Study Beyond 36 Months
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Stephen Lee, Professor and Chief, The University of Hong Kong
Other Study IDs: UW 14-456 (IRB HKU)
Record Dates: First submitted 2014-09-23; First posted 2014-10-13 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: Coronary Restenosis
Keywords: Safety and efficacy; Combo stent; Late loss thrombosis; Late loss catch up
MeSH Terms: conditions — Coronary Restenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- EGO-COMBO group: Previously enrolled into EGO-COMBO Pilot study and with combo stent
  Interventions: Other: EGO-COMBO group

INTERVENTIONS:
Other: EGO-COMBO group — Assess the safety and effectiveness of Combo stent

SUMMARY:
In this study, the safety and efficacy of COMBO TM stent beyond 36 months are assessed, in particular the occurrence of late stent thrombosis and late loss catch-up (restenosis).

DETAILED DESCRIPTION:
The Genous Stent (the EPC Capture R-stent, OrbusNeich Medical Inc., Fort Lauderdale, FL) is commercially available and has been used extensively in standard coronary intervention in the treatment of more than 200 patients with critical coronary stenoses at Queen Mary Hospital. The COMBO Stent (OrbusNeich Medical Inc., Fort Lauderdale, FL) is an improved version of the Genous Stent and is now widely available for clinical use in all Hong Kong hospitals. To date, more than 300 patients in Queen Mary Hospital have received the COMBO stent as treatment for their coronary artery disease, and all of them remained stable clinically.

The Genous Stent is a bio-engineered 316L stainless steel coronary stent with a biocompatible coating having specific CD34 antibody on the inner surface. CD34 is a surface antigen present on circulating endothelial progenitor cell (EPC). It will be bonded to the CD34 antibody, resulting in capturing of the EPC onto the stent surface and differentiation into endothelial layer. Animal model has demonstrated that a functional endothelial layer could be formed as soon as 24 to 48 hours after Genous stent implantation (1). The HEALING-FIM registry has shown that Genous stent is clinically safe and effective in the treatment of coronary stenosis (2). Recent reports have further confirmed its efficacy in patients with acute coronary syndrome requiring urgent revascularization (3,4).

The COMBO Stent is an improved version of the Genous Stent. The stent delivers a drug called sirolimus to the treated coronary blood vessel. This stent also incorporates a CD34 antibody coating that is designed to promote the healing of the treated coronary artery by catching endothelial progenitor cells from circulating blood as they pass through the stent. These cells are pro-healing and will help the blood vessel wall to heal over the stent more quickly and restore normal tissue function in the stented area. The combination of these two technologies in this new Combo stent is expected to produce even better clinical results, which are published in the REMEDEE Study.

Pre-clinical animal study has already shown the Combo Stent promoted endothelialization and reduced neointima formation, as assessed by both optical coherence tomography (OCT) and histopathology (5). However, such beneficial endothelial coverage as assessed by OCT has never been documented in human subjects, and has been addressed by previous study protocol: the EGO Study (IRB: UW 10-256), EGO-COMBO Pilot Study (UW 10-342) and EGO-COMBO angiographic extension study (UW 12-472). Queen Mary Hospital is currently the single cardiac centre worldwide with such vast experience in using the COMBO stent for percutaneous coronary intervention, together with intracoronary OCT to profile the stent's healing progress and subsequent neo-intimal growth and behaviour.

This current study protocol serves as an extension study to evaluate the long term clinical safety and efficacy of COMBO stent beyond 36 months post-implantation.

This is a single centre observational study to assess the safety and effectiveness clinical endpoints of COMBO TM stent beyond 36 months. Clinical notes for all subjects that previously participated in EGO-COMBO Pilot Study (UW 10-342) will be reviewed for clinical end points according to the definition of Academic Research Consortium and angina symptoms will be classified with Canadian Cardiovascular Society Angina Classification.

ELIGIBILITY:
Inclusion Criteria:

* Patient previously participated in EGO-COMBO Pilot Study (UW 10-342)

Exclusion Criteria:

* Patient not previously participated in EGO-COMBO Pilot Study (UW 10-342)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a single centre observational study to assess the safety and effectiveness clinical endpoints of COMBO TM stent beyond 36 months. Clinical notes for all subjects that previously participated in EGO-COMBO Pilot Study (UW 10-342) will be reviewed for clinical end points according to the definition of Academic Research Consortium and angina symptoms will be classified with Canadian Cardiovascular Society Angina Classification.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2014-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Composite Major Adverse Cardiac Events (MACE) | beyond 36 months

SECONDARY OUTCOMES:
All-cause mortality | beyond 36 months
Myocardial infarction | beyond 36 months
Target Lesion Revascularization | beyond 36 months
Angina Class | beyond 36 months
Target Vessel Failure | beyond 36 months
Cardiac Death | beyond 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Wai Luen Stephen LEE, MD, Principal Investigator — The Univeristy of Hong Kong
Locations (1):
- Department of Medicine, Queen Mary Hospital, The University of Hong Kong, Hong Kong, Hong Kong, China

REFERENCES:
- [Result] Prati F, Cera M, Ramazzotti V, Imola F, Giudice R, Albertucci M. Safety and feasibility of a new non-occlusive technique for facilitated intracoronary optical coherence tomography (OCT) acquisition in various clinical and anatomical scenarios. EuroIntervention. 2007 Nov;3(3):365-70. doi: 10.4244/eijv3i3a66. PMID 19737719
- [Result] Haude M, Lee SW, Worthley SG, Silber S, Verheye S, Erbs S, Rosli MA, Botelho R, Meredith I, Sim KH, Stella PR, Tan HC, Whitbourn R, Thambar S, Abizaid A, Koh TH, Den Heijer P, Parise H, Cristea E, Maehara A, Mehran R. The REMEDEE trial: a randomized comparison of a combination sirolimus-eluting endothelial progenitor cell capture stent with a paclitaxel-eluting stent. JACC Cardiovasc Interv. 2013 Apr;6(4):334-43. doi: 10.1016/j.jcin.2012.10.018. Epub 2013 Mar 20. PMID 23523459
- [Result] Yamaguchi T, Terashima M, Akasaka T, Hayashi T, Mizuno K, Muramatsu T, Nakamura M, Nakamura S, Saito S, Takano M, Takayama T, Yoshikawa J, Suzuki T. Safety and feasibility of an intravascular optical coherence tomography image wire system in the clinical setting. Am J Cardiol. 2008 Mar 1;101(5):562-7. doi: 10.1016/j.amjcard.2007.09.116. Epub 2008 Jan 10. PMID 18307999
- [Result] Granada JF, Inami S, Aboodi MS, Tellez A, Milewski K, Wallace-Bradley D, Parker S, Rowland S, Nakazawa G, Vorpahl M, Kolodgie FD, Kaluza GL, Leon MB, Virmani R. Development of a novel prohealing stent designed to deliver sirolimus from a biodegradable abluminal matrix. Circ Cardiovasc Interv. 2010 Jun 1;3(3):257-66. doi: 10.1161/CIRCINTERVENTIONS.109.919936. Epub 2010 May 4. PMID 20442358
- [Result] Co M, Tay E, Lee CH, Poh KK, Low A, Lim J, Lim IH, Lim YT, Tan HC. Use of endothelial progenitor cell capture stent (Genous Bio-Engineered R Stent) during primary percutaneous coronary intervention in acute myocardial infarction: intermediate- to long-term clinical follow-up. Am Heart J. 2008 Jan;155(1):128-32. doi: 10.1016/j.ahj.2007.08.031. Epub 2007 Nov 26. PMID 18082503
- [Result] Cutlip DE, Windecker S, Mehran R, Boam A, Cohen DJ, van Es GA, Steg PG, Morel MA, Mauri L, Vranckx P, McFadden E, Lansky A, Hamon M, Krucoff MW, Serruys PW; Academic Research Consortium. Clinical end points in coronary stent trials: a case for standardized definitions. Circulation. 2007 May 1;115(17):2344-51. doi: 10.1161/CIRCULATIONAHA.106.685313. PMID 17470709
- [Result] Aoki J, Serruys PW, van Beusekom H, Ong AT, McFadden EP, Sianos G, van der Giessen WJ, Regar E, de Feyter PJ, Davis HR, Rowland S, Kutryk MJ. Endothelial progenitor cell capture by stents coated with antibody against CD34: the HEALING-FIM (Healthy Endothelial Accelerated Lining Inhibits Neointimal Growth-First In Man) Registry. J Am Coll Cardiol. 2005 May 17;45(10):1574-9. doi: 10.1016/j.jacc.2005.01.048. PMID 15893169
- [Derived] Lee SW, Lam SC, Tam FC, Chan KK, Shea CP, Kong SL, Wong AY, Yung A, Zhang LW, Tse HF, Wu KK, Chan R, Haude M, Mehran R, Mintz GS, Maehara A. Evaluation of Early Healing Profile and Neointimal Transformation Over 24 Months Using Longitudinal Sequential Optical Coherence Tomography Assessments and 3-Year Clinical Results of the New Dual-Therapy Endothelial Progenitor Cell Capturing Sirolimus-Eluting Combo Stent: The EGO-Combo Study. Circ Cardiovasc Interv. 2016 Jul;9(7):e003469. doi: 10.1161/CIRCINTERVENTIONS.115.003469. PMID 27418609